CLINICAL TRIAL: NCT02288819
Title: Diuretic Efficiency in Patients With Stable Heart Failure: Ion Excretion Capacity of the Kidneys (DIPSTICK) Study
Brief Title: Spot Urinary Analysis to Assess Loop Diuretic Efficiency in Stable Heart Failure
Acronym: DIPSTICK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment and a lack of funding to complete further follow-up
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Mullens, MD PhD, Prof. Dr., Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOL-DIPSTICK
Record Dates: First submitted 2014-10-23; First posted 2014-11-11 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: loop diuretics; heart failure; natriuresis; urinary analysis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Loop diuretic downtitration (Experimental): Scheduled downtitration of maintenance loop diuretic dose while monitoring weight
  Interventions: Device: Weight monitoring; Drug: Loop diuretic downtitration

INTERVENTIONS:
Device: Weight monitoring — The body weight of patients is measured each morning in identical conditions on the same balance during 7 days
Drug: Loop diuretic downtitration — The patient's total daily maintenance dose of loop diuretics is downtitrated during 7 consecutive days.
  In case of a total daily maintenance dose ≤40 mg furosemide OR ≤1 mg bumetanide OR ≤20 mg torsemide, the loop diuretic is completely stopped.
  In case of a total daily maintenance dose >40 mg furosemide OR >1 mg bumetanide OR >20 mg torsemide, the loop diuretic dose is halved.

SUMMARY:
The primary objective of this study is to assess whether the urinary sodium/creatinine or chloride/creatinine ratio might predict successful downtitration of loop diuretics in patients with stable heart failure without clinical signs of volume overload. In addition, this study will provide information on loop diuretic efficiency and urinary electrolyte composition after intake of diuretics in stable outpatients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a left ventricular ejection fraction <40% or has been previously hospitalized with a primary diagnosis of heart failure
* Patient receives a daily maintenance dose of loop diuretics

Exclusion Criteria:

* Patient was hospitalized for heart failure <3 months before study inclusion
* The maintenance dose of loop diuretics was changed <3 months before study inclusion
* The maintenance dose of renin-angiotensin-aldosterone system blockers or beta-blocker medication was changed <3 months before study inclusion
* Cardiac resynchronization therapy (CRT) was initiated <3 months before study inclusion
* At the moment of inclusion, the patient has either one of the following signs of volume overload: lower leg edema +2/4, ascites, lung congestion
* Patient is not able to measure his/her weight safely and correct at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Mullens, M.D. Ph.D., Principal Investigator — Ziekenhuis Oost-Limburg; Frederik H Verbrugge, M.D. Ph.D., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martens P, Verbrugge FH, Boonen L, Nijst P, Dupont M, Mullens W. Value of routine investigations to predict loop diuretic down-titration success in stable heart failure. Int J Cardiol. 2018 Jan 1;250:171-175. doi: 10.1016/j.ijcard.2017.10.018. Epub 2017 Oct 6. PMID 29056238
- [Result] Verbrugge FH, Martens P, Boonen L, Nijst P, Verhaert D, Noyens P, De Vusser P, Dupont M, Tang WHW, Mullens W. Loop diuretic down-titration in stable chronic heart failure is often achievable, especially when urinary chloride concentration is low. Acta Cardiol. 2018 Aug;73(4):335-341. doi: 10.1080/00015385.2017.1385152. Epub 2017 Oct 3. PMID 28971753
- [Result] Boonen L, Verbrugge FH, Nijst P, Noyens P, De Vusser P, Verhaert D, Van Lierde J, Vrolix M, Dupont M, Mullens W. Subclinical volume overload in stable outpatients with chronic heart failure. Acta Cardiol. 2016 Jun;71(3):299-307. doi: 10.2143/AC.71.3.3152090. No abstract available. PMID 27594125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient cardiology clinic of a single tertiary centre (Ziekenhuis Oost-Limburg, Genk, Belgium) between December, 2014, and February, 2016.
Groups:
- Loop Diuretic Downtitration: Scheduled downtitration of maintenance loop diuretic dose while monitoring weight
  Weight monitoring: The body weight of patients is measured each morning in identical conditions on the same balance during 7 days
  Loop diuretic downtitration: The patient's total daily maintenance dose of loop diuretics is downtitrated during 7 consecutive days.
  In case of a total daily maintenance dose ≤40 mg furosemide OR ≤1 mg bumetanide OR ≤20 mg torsemide, the loop diuretic is completely stopped.
  In case of a total daily maintenance dose >40 mg furosemide OR >1 mg bumetanide OR >20 mg torsemide, the loop diuretic dose is halved.
Period: Overall Study
Arm/Group | Loop Diuretic Downtitration
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [61 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Downtitration of Loop Diuretics (no Weight Increase >1,5 kg)
Description: After baseline evaluation, loop diuretics are temporarily downtitrated or stopped for 7 consecutive days. The patient is instructed to measure his/her weight in the morning of these days, immediately after waking up, on the same balance. In case of weight increase >1,5 kg, the original dose of diuretics is restored. To check this, patients are contacted by phone after 3 and 7 days. If the patient has not gained >1,5 kg of weight after 7 days, loop diuretics are considered to be successfully downtitrated.
Time Frame: 7 days after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 50
Participants | 37

2. Secondary Outcome: All-cause Mortality
Time Frame: 30 days after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 50
Participants | 1

3. Secondary Outcome: Number of Participants Rehospitalized for Heart Failure
Description: Unplanned hospital admission for symptoms of congestion and/or low output heart failure requiring either intravenous therapy and/or increase of oral diuretics.
Time Frame: 30 days after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 50
Participants | 1

4. Secondary Outcome: Number of Participants Requiring a Dose Increase in Loop Diuretics
Description: Dose increase of oral maintenance therapy with loop diuretics compared to the final dose achieved in the study 7 days after baseline.
Time Frame: 30 days after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 50
Participants | 1

5. Secondary Outcome: Weight Change
Description: Weight change [kg] 7 days after baseline compared to baseline weight.
Time Frame: 7 days after baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 50
kg | 0.502 (1.101)

6. Other Pre Specified Outcome: Weight Change
Description: Weight change [kg] 30 days after baseline compared to weight 7 days after baseline (after achieving the final dose of loop diuretics).
Time Frame: 30 days after baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 43
kg | -0.261 (1.391)

7. Other Pre Specified Outcome: Self-reported Orthopnea
Description: The patient is contacted by phone 30 days after baseline and asked for self-reported orthopnea.
Time Frame: 30 days after baseline
Population: 1 patient who died before the 30-day follow-up could not be assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 49
Participants | 5

8. Other Pre Specified Outcome: Self-reported Lower Leg Edema
Description: The patient is contacted by phone 30 days after baseline and asked for self-reported presence of lower leg edema.
Time Frame: 30 days after baseline
Population: 1 patient who died before the 30-day follow-up could not be assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 49
Participants | 1

9. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Class
Description: NYHA class is a semi-quantitative measurement of functional capacity on a scale from 1 to 4:
  1. No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  2. Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  3. Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  4. Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  For the purpose of this outcome parameter, the patient is contacted by phone 30 days after baseline and NYHA functional class is assessed by a study investigator.
Time Frame: 30 days after baseline
Population: 1 patient who died before the 30-day follow-up could not be assessed
Measure: Mean (Standard Deviation); unit: units on a scale from 1 to 4
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 49
units on a scale from 1 to 4 | 1.41 (0.57)

10. Other Pre Specified Outcome: All-cause Mortality
Time Frame: 6 months after baseline
Population: The study was terminated after every participant reached the 30-day follow-up point because of slow recruitment and a lack of funding to complete further follow-up
Arm/Group | Loop Diuretic Downtitration
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Rehospitalization for Heart Failure
Description: as for outcome 3
Time Frame: 6 months after baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Dose Increase of Loop Diuretics
Description: as for outcome 4
Time Frame: 6 months after baseline
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Weight Change
Description: Weight change [kg] 7 days after baseline compared to baseline weight.
Time Frame: 7 days after baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Self-reported Orthopnea
Description: The patient is contacted by phone 30 days after baseline and asked for self-reported orthopnea.
Time Frame: 30 days after baseline
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Self-reported Lower Leg Edema
Description: The patient is contacted by phone 30 days after baseline and asked for self-reported presence of lower leg edema.
Time Frame: 30 days after baseline
Reporting Status: Not Posted

16. Other Pre Specified Outcome: NYHA Functional Class
Description: The patient is contacted by phone 30 days after baseline and NYHA functional class is assessed by a study investigator.
Time Frame: 30 days after baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Loop Diuretic Downtitration
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 1/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loop Diuretic Downtitration (N=50)
Heart failure readmission (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No